CLINICAL TRIAL: NCT00886431
Title: A Double Blinded, Randomised Controlled Trial Comparing the Effectiveness of Vitrification to Slow Cooling in Cryopreserving Human Preimplantation Embryos
Brief Title: Vitrification Versus Slow Cooling of Human Cleavage Stage Embryos
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, Prof. dr. B Fauser, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vitrification study; CCMO NL23499.000.08; METC 08/183
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Infertility
Keywords: IVF; embryo cryopreservation; vitrification; slow cooling; slow freezing; surplus embryos; Human Reproduction
MeSH Terms: conditions — Infertility | interventions — Vitrification

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrification (Experimental): The embryos of patients allocated to this arm will be cryopreserved by vitrification.
  Interventions: Other: embryo vitrification
- Slow cooling (No Intervention): The embryos of patients allocated to this arm will be cryopreserved by the slow cooling method, which is the standard method (=no intervention)

INTERVENTIONS:
Other: embryo vitrification — Ultra rapid cooling of embryos by immersion in liquid nitrogen. The formation of potentially damaging ice crystals is prevented by briefly incubating the embryos in high concentrations of a mix of cryoprotectants.
  Other Names: vitrification; high security vitrification straws
  Arms: Vitrification

SUMMARY:
Human embryos can be preserved for later transfers by freezing. Traditionally the slow cooling method has been used. About 70% of the embryos remain fully intact after thawing. However, the remaining 30% of the embryos become (partially) damaged, and this freezing damage reduces their chance to implant. Recently an ultra rapid freezing method, called vitrification has been developed. During vitrification no damaging ice crystals are formed and the embryo freezes in a glass like state.

It appears that the freezing damage is reduced when embryos are vitrified. Observational studies in humans indicate that embryos are successfully preserved by vitrification, as indicated by promising pregnancy rates following thawing. However, the effectiveness of vitrification in relation to slow cooling with respect to pregnancy rates has so far not been evaluated by a randomised, controlled trial. The aim of this study is to investigate whether vitrification significantly improves embryo survival and ongoing pregnancy rates when compared to embryos frozen by slow cooling.

DETAILED DESCRIPTION:
time of allocation: following embryo selection

type of embryos: cleavage stage -, morula stage or early blastocyst stage embryo (day3 - day4 after oocyte collection)

cryoprotectants: sucrose, dimethylsulfoxide, ethyleneglycol

vitrification storage device: high security vitrification straws

ELIGIBILITY:
Inclusion Criteria:

* female patient age 35 years or less
* embryos are obtained by in vitro fertilization (IVF) or intra cytoplasmatic spermatozoon injection (ICSI)
* single embryo transfer
* 1rst IVF/ICSI treatment with an embryo transfer
* availability of cryopreservable embryos

Exclusion Criteria:

* female patient age is 36 years or older
* participants of oocyte donation program
* participants of percutaneous spermatozoon aspiration (PESA) program
* couples with a finite source of spermatozoa
* absence of cryopreservable embryos

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The percent change of the ongoing pregnancy rate per patient/couple who use their thawed embryos (following a fesh embryo transfer which did not result in an ongoing pregnancy) from baseline (slow cooling) to end point (vitrification). | ongoing pregnancy is established 10 weeks following the transfer of a frozen embryo

SECONDARY OUTCOMES:
post-thaw embryo survival rate | 1 hour after thawing
ongoing pregnancy rate per patient using their thawed embryos (independent of whether they became pregnant following a fresh embryo transfer or not | 10 weeks following transfer of frozen thawed embryo
implantation rate per thawed embryo | 10 weeks after transfer of thawed embryo
implantation rate per transferred thawed embryo | 10 weeks after transfer of thawed embryo
cumulative implantation rate per cryopreservation | 10 weeks after thawed embryo transfer
ongoing pregnancy rate per frozen-thaw cycle | 10 weeks following thawed embryo transfer
average number of frozen-thawed cycles per patient | is variable
post thaw development (categorial) per thawed embryo | 24 hours following thawing
average number of cryo-thaw cycles to ongoing pregnancy | variable, up to 3 years
average number of thawed embryos to ongoing implantation | variable, up to 3 years
Life birth rate | 9 month after pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Bart C Fauser, Prof.,MD,PhD, Principal Investigator — UMC Utrecht
Locations (2):
- Academic Hospital of Brussels, Brussels, Belgium
- University Medical Center of Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Boonkusol D, Gal AB, Bodo S, Gorhony B, Kitiyanant Y, Dinnyes A. Gene expression profiles and in vitro development following vitrification of pronuclear and 8-cell stage mouse embryos. Mol Reprod Dev. 2006 Jun;73(6):700-8. doi: 10.1002/mrd.20450. PMID 16541460
- [Background] Burns WN, Gaudet TW, Martin MB, Leal YR, Schoen H, Eddy CA, Schenken RS. Survival of cryopreservation and thawing with all blastomeres intact identifies multicell embryos with superior frozen embryo transfer outcome. Fertil Steril. 1999 Sep;72(3):527-32. doi: 10.1016/s0015-0282(99)00280-0. PMID 10519629
- [Background] Desai N, Blackmon H, Szeptycki J, Goldfarb J. Cryoloop vitrification of human day 3 cleavage-stage embryos: post-vitrification development, pregnancy outcomes and live births. Reprod Biomed Online. 2007 Feb;14(2):208-13. doi: 10.1016/s1472-6483(10)60789-4. PMID 17298725
- [Background] Edgar DH, Bourne H, Speirs AL, McBain JC. A quantitative analysis of the impact of cryopreservation on the implantation potential of human early cleavage stage embryos. Hum Reprod. 2000 Jan;15(1):175-9. doi: 10.1093/humrep/15.1.175. PMID 10611209
- [Background] Kasai M, Mukaida T. Cryopreservation of animal and human embryos by vitrification. Reprod Biomed Online. 2004 Aug;9(2):164-70. doi: 10.1016/s1472-6483(10)62125-6. PMID 15333245
- [Background] Mukaida T, Nakamura S, Tomiyama T, Wada S, Kasai M, Takahashi K. Successful birth after transfer of vitrified human blastocysts with use of a cryoloop containerless technique. Fertil Steril. 2001 Sep;76(3):618-20. doi: 10.1016/s0015-0282(01)01968-9. PMID 11532492
- [Background] Rama Raju GA, Haranath GB, Krishna KM, Prakash GJ, Madan K. Vitrification of human 8-cell embryos, a modified protocol for better pregnancy rates. Reprod Biomed Online. 2005 Oct;11(4):434-7. doi: 10.1016/s1472-6483(10)61135-2. PMID 16274602
- [Background] Salumets A, Suikkari AM, Makinen S, Karro H, Roos A, Tuuri T. Frozen embryo transfers: implications of clinical and embryological factors on the pregnancy outcome. Hum Reprod. 2006 Sep;21(9):2368-74. doi: 10.1093/humrep/del151. Epub 2006 May 9. PMID 16684837
- [Background] Sheehan CB, Lane M, Gardner DK. The CryoLoop facilitates re-vitrification of embryos at four successive stages of development without impairing embryo growth. Hum Reprod. 2006 Nov;21(11):2978-84. doi: 10.1093/humrep/del253. Epub 2006 Sep 1. PMID 16950825
- [Background] Stehlik E, Stehlik J, Katayama KP, Kuwayama M, Jambor V, Brohammer R, Kato O. Vitrification demonstrates significant improvement versus slow freezing of human blastocysts. Reprod Biomed Online. 2005 Jul;11(1):53-7. doi: 10.1016/s1472-6483(10)61298-9. PMID 16102287
- [Background] Takahashi K, Mukaida T, Goto T, Oka C. Perinatal outcome of blastocyst transfer with vitrification using cryoloop: a 4-year follow-up study. Fertil Steril. 2005 Jul;84(1):88-92. doi: 10.1016/j.fertnstert.2004.12.051. PMID 16009162
- [Background] Al-Hasani S, Ozmen B, Koutlaki N, Schoepper B, Diedrich K, Schultze-Mosgau A. Three years of routine vitrification of human zygotes: is it still fair to advocate slow-rate freezing? Reprod Biomed Online. 2007 Mar;14(3):288-93. doi: 10.1016/s1472-6483(10)60869-3. PMID 17359578
- [Background] Liebermann J, Tucker MJ. Comparison of vitrification and conventional cryopreservation of day 5 and day 6 blastocysts during clinical application. Fertil Steril. 2006 Jul;86(1):20-6. doi: 10.1016/j.fertnstert.2006.01.029. Epub 2006 Jun 8. PMID 16762345
- [Background] Yokota Y, Sato S, Yokota M, Yokota H, Araki Y. Birth of a healthy baby following vitrification of human blastocysts. Fertil Steril. 2001 May;75(5):1027-9. doi: 10.1016/s0015-0282(01)01685-5. PMID 11334922